CLINICAL TRIAL: NCT00350519
Title: An Open Label, Multicenter, Randomized, Controlled Study to Evaluate Efficacy and Safety of PROCRIT in Subjects Undergoing Elective Major Abdominal and/or Pelvic Surgery
Brief Title: The Safety and Effectiveness of PROCRIT (Epoetin Alfa) in Patients Undergoing Elective Major Abdominal and/or Pelvic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped due to slow enrollment
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012460; EPOSUR4005 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Results first posted 2009-05-06 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Hemostasis, Surgical
Keywords: Hemostasis, Surgical; Epoetin alfa; Surgery; Abdomen; Pelvis; PROCRIT; pRBC; Blood transfusion; Packed red blood cell transfusion
MeSH Terms: interventions — Epoetin Alfa; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PROCRIT (epoetin alfa) (Experimental): Participants will receive PROCRIT (epoetin alfa).
  Interventions: Drug: Epoetin alfa
- STANDARD THERAPY (Experimental): Participants will receive standard of care.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Epoetin alfa — Participants will receive epoetin alfa 300 IU/kg once daily subcutaneously for 10 days prior to surgery, on the day of surgery, and for four days after surgery.
  Other Names: PROCRIT
  Arms: PROCRIT (epoetin alfa)
Drug: Standard of Care — Participants will receive standard of care based on the Institution's treatment policy.
  Arms: STANDARD THERAPY

SUMMARY:
The primary purpose of the study is to compare the effect of perioperative (the time period describing the duration of a participants surgical procedure) administration of PROCRIT to that of Standard of Care (SOC) on the proportion of participants receiving pRBC (packed red blood cells) transfusions (from the day of surgery to the day of hospital discharge) in participants undergoing elective major abdominal and/or pelvic surgery. Standard of Care is defined as the treatment of participants according to the hospital or institution's policy, but where participants will not receive PROCRIT (Epoetin alfa) or any other erythropoiesis-stimulating agents (ESAs) (agents that stimulate the production of red blood cells in the bone marrow).

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), parallel-arm (each group of participants will be treated at the same time), open-label (all people know the identity of the intervention), multicenter study. The study consists of screening phase of 21 days, treatment phase of 15 days, follow-up phase of 28 days. Approximately 110 participants undergoing elective major abdominal and/or pelvic surgery will be enrolled. During the Treatment Phase, eligible participants will be randomly assigned (participants are assigned to a treatment group based on chance) in a 1:1 ratio to either PROCRIT (Epoetin alfa) or the Standard of Care (SOC) group that will not receive any erythropoiesis-stimulating agents (ESAs). Participants will undergo surgery during the Treatment Phase. After surgery, all participants will stay in the study for 4 days (or until hospital discharge) and followed for an additional 28 days (Follow-up Phase). Safety evaluations will include assessment of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination which will be monitored throughout the study. The duration of the study for each participant will be approximately 64 days.

ELIGIBILITY:
Inclusion Criteria: - Scheduled to undergo elective major abdominal and/or pelvic surgery with anticipated significant perioperative ((the time period describing the duration of a participants surgical procedure) blood loss (eg, greater than 500 cc and at increased risk for blood transfusion) - Hemoglobin greater than 10 g/dL and less than or equal to 13 g/dL at screening (Day -13 [13 days prior to surgery] to Day -11) and baseline (Day -10) - Patients with reproductive potential and their partners must practice an effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, partner sterilization) before entry and throughout the study - Female patients with reproductive potential must have a negative urine pregnancy test within 7 days of the first dose of PROCRIT - Adequate renal (kidney) and adequate hepatic (liver) function assessed within the 21-day screening period Exclusion Criteria: - No severe Congestive Heart Failure (New York Heart Association Class IV) - No known severe stable or unstable coronary artery disease, or unstable angina - No history of deep venous thrombosis (DVT) or pulmonary embolus (PE) within 12 months before study entry (prior superficial thrombophlebitis is not an exclusion criterion) - No history of cerebrovascular accident (CVA), transient ischemic attack (TIA), Acute coronary syndrome (unstable Angina, myocardial Infarction), or other arterial thrombosis within 6 months before study entry - Not anticipated to donate perioperative autologous blood or receive transfusions within 21 days prior to baseline or to have greater than 6 transfusions perioperatively - No prior treatment with PROCRIT or any erythropoiesis-stimulating agents (ESAs) within the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 participants were enrolled in the study. 18 participants were randomly assigned to the epoetin alfa group and 19 were randomly assigned to the Standard therapy group.
Groups:
- PROCRIT (Epoetin Alfa): Participants received epoetin alfa 300 IU/kg subcutaneously once daily for 10 days, prior to surgery, on the day of surgery, and for four days after surgery
- STANDARD THERAPY: Participants received standard of care based on the Institution's treatment policy
Period: Overall Study
Arm/Group | PROCRIT (Epoetin Alfa) | STANDARD THERAPY
Started | 18 | 19
Completed | 14 | 13
Not Completed | 4 | 6
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PROCRIT (Epoetin Alfa) | STANDARD THERAPY | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 7 | 7 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 63.06 (16.17) | 61.42 (18.32) | 62.22 (17.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 5 | 9 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Black or Aftrican American | 0 | 5 | 5
  Other | 1 | 2 | 3
  White | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving pRBC (Packed Red Blood Cell) Transfusions
Time Frame: Day of surgery until hospital discharge
Population: ITT(intention to treat), No formal analysis was conducted due to early termination and small sample size
Measure: Number; unit: participants
Arm/Group | PROCRIT (Epoetin Alfa) | STANDARD THERAPY
Number analyzed (Participants) | 18 | 19
participants | 4 | 9

2. Secondary Outcome: Hemoglobin Change From Baseline to End of Study
Description: End of Study Hemoglobin minus baseline Hemoglobin
Time Frame: Baseline (Day-10) to end of study (Day 32)
Population: All Subjects, No formal analysis was conducted due to early termination and small sample size
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | PROCRIT (Epoetin Alfa) | STANDARD THERAPY
Number analyzed (Participants) | 13 | 13
g/dL | 0.98 (1.39) | 0.33 (2.06)

3. Secondary Outcome: Number of pRBC Units Transfused During Study
Time Frame: Baseline (Day -10) to end of study (Day 32)
Population: ITT, No formal analysis was conducted due to early termination and small sample size
Measure: Mean (Standard Deviation); unit: units
Arm/Group | PROCRIT (Epoetin Alfa) | STANDARD THERAPY
Number analyzed (Participants) | 4 | 9
units | 3.5 (3.00) | 6.11 (7.98)

4. Secondary Outcome: Hospital Length of Stay
Time Frame: Surgery to hospital discharge
Population: ITT, No formal analysis was conducted due to early termination and small sample size
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PROCRIT (Epoetin Alfa) | STANDARD THERAPY
Number analyzed (Participants) | 17 | 16
days | 7.94 (5.17) | 12.56 (12.30)

ADVERSE EVENTS:
Time Frame: 64 days
Arm/Group | PROCRIT (Epoetin Alfa) | STANDARD THERAPY
Serious Adverse Events (participants affected / at risk) | 5/18 | 8/19
Other Adverse Events (participants affected / at risk) | 18/18 | 13/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PROCRIT (Epoetin Alfa) (N=18) | STANDARD THERAPY (N=19)
Abdominal abscess (Infections and infestations) | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level below therapurtic (Investigations) | 0 | 1
International normalized ratio increased (Investigations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2
Hypergylcaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PROCRIT (Epoetin Alfa) (N=18) | STANDARD THERAPY (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 6
Pancreatic fistula (Gastrointestinal disorders) | 1 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Asthenia (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 7
Application site infection (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 3
Procedural hypotension (Injury, poisoning and procedural complications) | 3 | 5
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Blood potassium decreased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Prothrombin level increased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 0 | 2
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Wound drainage (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 5

LIMITATIONS AND CAVEATS:
No formal analysis was conducted due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days